CLINICAL TRIAL: NCT03202238
Title: TenTaTorch: Venepuncture Made Easy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2018/01266
Record Dates: First submitted 2017-04-16; First posted 2017-06-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Vein Collapse; Vein Thrombosis; Vein; Tortuous; Vein Disease
MeSH Terms: conditions — Venous Thrombosis | interventions — Congresses as Topic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional (Active Comparator): Venepuncture without the use of any venepuncture assistive device
  Interventions: Other: Conventional
- Veinlite (Active Comparator): Commercial transilluminator device that allows veins to show up as a silhouette among surrounding soft tissue
  Interventions: Device: Veinlite
- TenTaTorch (Experimental): Transilluminator device that allows veins to show up as a silhouette among surrounding soft tissue
  Interventions: Device: TenTaTorch

INTERVENTIONS:
Other: Conventional — Conventional venepuncture without use of any venepuncture assistive device.
  Arms: Conventional
Device: Veinlite — Commercial transilluminator device that allows veins to show up as a silhouette among surrounding soft tissue
  Arms: Veinlite
Device: TenTaTorch — Transilluminator device that allows veins to show up as a silhouette among surrounding soft tissue
  Arms: TenTaTorch

SUMMARY:
Venepuncture can be challenging, especially in patients with co-morbidities that predispose them to have inaccessible veins. Multiple unsuccessful venepuncture attempts compromise patient care. It causes pain, delays in obtaining blood samples for investigations and instituting intra-venous treatment.

Venepuncture assistive devices (VAD) include ultrasonography, and devices that utilize infra-red or transillumination. These are expensive, not widely available, and have not been rigorously proven to be effective. We have previously performed a preliminary study using an ordinary pen-torch for transillumination showed promising results. 95% of patients with known difficult venous access required two or less attempts for successful cannulation. It costs 35 times cheaper compared to the cheapest VAD in the market. The concept is promising but the technique cumbersome.

Building upon the concept of transillumination, the aim of this study is to develop an idiot-proof cost-effective pocket-sized VAD (TenTaTorch) to improve venepuncture success. A randomized controlled trial (RCT) will be conducted to determine its safety and efficacy. The TenTaTorch prototype will be modelled using Computer-Aided Design (Inventor®, Autodesk®, California, USA) and fabricated using 3D-printing, with silicon casting. Compared to existing VADs, TenTaTorch consists of finger-mounted LED light sources that allows greater manoeuvrability during transillumination.

We include adult patients aged 21 to 100 with difficult venous access (history of ≥3 consecutive attempts required for successful cannulation during the current admission) requiring non-emergent venepuncture in the RCT. Each patient undergoes venepuncture over the upper-limb using one of the following: Conventional Venepuncture without aid (Control 1); Veinlite® EMS (TransLite®, Texas, USA) (Control 2), a commercial transillumination device; our device TenTaTorch (Experimental Group).

Outcome measures include: successful cannulation within 2 attempts; duration of venepuncture; subjective user feedback. Fisher's exact and Kruskal-Wallis tests will be performed.

DETAILED DESCRIPTION:
This is a prospective randomized controlled trial. Patients with a history of difficult venepuncture who agreed to be enter into the study will be randomized into one of three groups using a sealed envelope system: Conventional Venepuncture without aid (Control 1); Veinlite® EMS (TransLite®, Texas, USA) (Control 2), a commercial transillumination device; our device TenTaTorch (Experimental Group). Hemodynamically unstable patients are excluded. The nurse involved in the care of the patient will attempt venepuncture over the upper limb. A group of nurses will be recruited before the start of patient recruitment. A maximum of 4 times attempts is allowed, before escalation to a doctor/phlebotomist.

A standardized venepuncture technique using standardized instruments will be utilized. A tourniquet is applied (Braun® International, USA). Veins will be localized using one of the above techniques. Both Veinlite and TenTaTorch utilize the concept of transillumination. Placing it onto the skin will cause the outlines of the veins to show up. Once a suitable vein is localized, the vein is marked with a pen. The area of the skin to be cannulated is disinfected with an alcohol wipe (Webcol®, Covidien®, USA). For the setting of IV cannulation, a standardized IV cannula (ranging 18 to 25 gauge) is used (Introcan Safety®, Braun®, USA). Normal saline (PosiFlush® 3ml, BD®, USA) will be used for flushing the cannula after successful cannulation. For blood taking, a syringe (Terumo®, Philippines) ranging from 2ml to 20ml and a needle (ranging between 18 to 25 gauge) (Venofix®, Braun®, USA) will be used. All instruments needed for venepuncture, including 4 IV cannula or 4 needles should be by the patient's bedside prior to the start of each venepuncture attempt. Duration of the procedure will be recorded using a stop watch. This is defined as the time (in minutes) from the start of attempt to localize a vein to its successful cannulation. Successful cannulation is defined either as the ability to flush 2ml of normal saline into the IV cannula or the ability to draw 2ml of blood from the vein. A post-procedure questionnaire will be filled up by the nurses after the attempt at venepuncture.

Outcome data include: number of attempts and duration needed for successful venepuncture. Patient data include: age, sex, race, body-mass index, history of intra-venous drug abuse, and renal function. Nurses who consent to join the study will be required to participate in a pre- trial tutorial which is estimated to last for 1 hour. During the tutorial, techniques of locating veins using TenTaTorch and by using the Veinlite® device will be taught. A standardized technique of venepuncture will also be taught. Tutorial will be in the form of slide- show presentation and hands-on training. During the hands-on training, nurses will attempt to identify veins on fellow trainees using both TenTaTorch and Veinlite®.

ELIGIBILITY:
Inclusion Criteria:

* Patients with difficult venous access: Patients who have a history of 3 or more venepuncture attempts required for successful cannulation

Exclusion Criteria:

* Patients who require emergency blood sampling
* Patients who require emergency insertion of intra-venous cannula
* Patients who are haemodynamically unstable

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-09-29 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-10-05 (Estimated)

PRIMARY OUTCOMES:
Number of attempts | Up to 1 day from the point of venepuncture attempt
  Number of venepuncture attempts required for successful vein cannulation

SECONDARY OUTCOMES:
Duration of venepuncture | Up to 1 day from the point of venepuncture attempt
  Duration required for successful vein cannulation

OTHER OUTCOMES:
Subjective user feedback | Up to 1 day from the point of venepuncture attempt
  User feedback on the ease of use of the device which would include information on the following:
  1. Ranking of the ease of use of different venepuncture assistive devices
  2. Evaluating the devices on the ease of use on a scale of 1 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Elijah Cai, MBBS, MRCS, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No